CLINICAL TRIAL: NCT06348251
Title: Evaluating a Digital Intervention for Binge Eating and Weight Management Among Adults With Food Insecurity
Brief Title: FoodSteps for Binge Eating & Food Insecurity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Andrea Graham, Associate Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00219612
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Binge Eating; Type 2 Diabetes; Food Insecurity
MeSH Terms: conditions — Bulimia; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral intervention (Other)
  Interventions: Behavioral: FoodSteps

INTERVENTIONS:
Behavioral: FoodSteps — Participants will get access to the FoodSteps digital intervention with coaching for 16 weeks and receive a weekly stipend benefit to aid with implementing health behavior changes

SUMMARY:
The purpose of this study is to conduct a pilot trial of a mobile intervention that targets binge eating and weight-related behaviors, to determine the feasibility, acceptability, and preliminary efficacy of the intervention among adults with recurrent binge eating, diabetes, and food insecurity.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or older
* Recurrent binge eating (≥12 episodes in the past 3 months)
* Type 2 diabetes mellitus
* Food insecure status (e.g. difficulty accessing food)
* Interested in losing weight and reducing binge eating
* Willing to use a mobile application
* Has a smartphone with Internet access and capacity for calls and text messaging
* Has a valid email address
* Not pregnant
* English-speaking

Exclusion Criteria:

* Diagnosis for which the study/intervention is not clinically indicated
* Currently receiving clinical services for weight management or binge eating
* Started or recently (within the past month) changed dosage of a medication for binge eating, weight management, or diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FoodSteps: Digital intervention with coaching for 16 weeks and a weekly stipend benefit
Period: Overall Study
Arm/Group | FoodSteps
Started | 31
Completed | 30
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | FoodSteps
Number analyzed (Participants) | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 9
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.45 (11.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 23
  Male | 7
  Not reported as male or female | 1

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Feasibility assessed by study recruitment and retention rates
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FoodSteps
Number analyzed (Participants) | 31
Participants | 30

2. Primary Outcome: Study Retention Rate
Description: Feasibility assessed by study recruitment and retention rates
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FoodSteps
Number analyzed (Participants) | 31
Participants
  Retained | 30
  Withdrew | 1

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | FoodSteps
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT06348251/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT06348251/SAP_001.pdf